CLINICAL TRIAL: NCT03142113
Title: A Retrospective Multicentric Belgian Observational Trial to Evaluate the Successfulness of Adalimumab Dose Escalation and De-escalation in Patients With Moderate-to-severe Ulcerative Colitis Treated With Adalimumab
Brief Title: Clinical Outcome After Escalation and De-escalation of Adalimumab in Real Life in Ulcerative Colitis
Acronym: CEDAR UC
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Belgian Inflammatory Bowel Disease Research and Development (BIRD) VZW (Other); Imelda Hospital, Bonheiden (Other); University of Liege (Other); Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other); AZ Delta (Other); Algemeen Ziekenhuis Maria Middelares (Other); University Hospital, Ghent (Other); General Hospital Groeninge (Other); Centre Hospitalier Universitaire UCLouvain Namur (Other); Université Catholique de Louvain (Other); Onze Lieve Vrouwziekenhuis Aalst (Other)
Responsible Party: Sponsor
Other Study IDs: S59663
Record Dates: First submitted 2016-10-26; First posted 2017-05-05 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Ulcerative Colitis
Keywords: optimization; adalimumab
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This retrospective multi-centric Belgian observational trial will involve all patients who have initiated adalimumab for moderate-to-severe ulcerative colitis prior to September 1st 2015 in a Belgian centre maintaining a prospective log of patients using biological therapy.

Only patients fulfilling all Belgian reimbursement criteria for adalimumab will be included, namely having failed mesalamine and steroids or thiopurine analogues for at least 3 months, or being intolerant to this therapy, and showing a total Mayo score of at least 6 with an endoscopic sub-score of at least 2.

Both short-term and long-term outcome of adalimumab therapy will be evaluated, focusing on the need and successfulness of adalimumab dose-escalation from 40mg every other week to 40mg every week, and dose de-escalation back to 40mg every other week.

DETAILED DESCRIPTION:
Adalimumab is approved for the treatment of moderate to severe ulcerative colitis after failure of aminosalicylates plus corticosteroids and/or immunomodulators.1-4 In the registration studies for adalimumab in ulcerative colitis prior anti-tumor necrosis factor (TNF) treatment was restricted; in ULTRA 1, prior anti-TNF treatment was an exclusion criterion,5 while in ULTRA 2, 40% of patients had been exposed to infliximab prior to start of adalimumab, but primary non-responders to infliximab were excluded.6 Open label real life studies have shown good responses to adalimumab in UC. However typically, these cohorts were small and most patients were anti-TNF naïve. One Italian open label study on 88 patients reported clinical remission rates of 28% and 43% at week 12 and year 1, respectively.7 No significant differences were observed between infliximab naïve and infliximab exposed UC patients. In a Belgian open label study of 73 patients previously failing infliximab, overall clinical response at week 12 and 52 were 75% and 52%, respectively.8 Adalimumab was continued without need for dose escalation throughout year 1 in 16 patients, 22 needed dose escalation and 35 discontinued treatment within 1 year. Prior response to infliximab and early serum concentrations correlated with response.

While data are available in Crohn's disease,9 real life data on adalimumab dose escalation and dose de-escalation are limited in ulcerative colitis. Similarly, factors associated with need and success of dose escalation and dose de-escalation later on are almost absent.

ELIGIBILITY:
Site Selection:

* Only Belgian sites are eligible
* Participating sites must maintain a patient log allowing a full coverage of patients eligible for this study
* Membership of the Belgian IBD Research and Development (BIRD) group is not mandatory
* Local investigator is willing and able to fill out a two page case report form (CRF) for each eligible patient in a two month period (deadline November 1st 2016)

Inclusion Criteria:

* Age at least 18 at initiation of adalimumab therapy
* Adalimumab initiated before September 1st 2015
* Established diagnosis of ulcerative colitis
* Having failed mesalamine and steroids or thiopurine analogues for at least 3 months, or being intolerant to this therapy (as described in the Belgian reimbursement criteria)
* Active ulcerative colitis as described in the Belgian reimbursement criteria, namely showing a total Mayo score of at least 6 with an endoscopic sub-score of at least 2

Exclusion Criteria:

* Subjects with Crohn's disease or inflammatory bowel disease (IBD) type unclassified
* Subjects previously treated with adalimumab
* Subjects treated with adalimumab for other reasons than moderate-to-severe ulcerative colitis, including extra-intestinal manifestations and pre-emptively switch from other biological therapies (i.e. while being in clinical remission)
* Subjects who underwent subtotal colectomy or proctocolectomy prior to adalimumab initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enrol all subjects who initiated adalimumab for moderate-to-severe ulcerative colitis before September 1st 2015 at 11 sites throughout Belgium. These 11 sites have pre-screened their database, and almost 300 patients seem eligible.
Sampling Method: Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
The need and success of adalimumab dose escalation from 40mg every other week to 40mg every week in patients with moderate-to-severe ulcerative colitis during adalimumab treatment | Through study completion, an average of 24 months
  The proportion of patients requiring dose-escalation from adalimumab 40mg every other week to 40mg every week and the success rate of this intervention.
  Success of dose-escalation is defined based on a positive physician global assessment and absence of blood on two consecutive visits at least 3 months apart from each other. Of note: patients requiring a second intervention later on (addition of any type of steroids, addition of any immunomodulatory drug or optimization to off-label adalimumab 80 mg every week) will be regarded as failure (treatment optimization based on trough level monitoring or biomarkers alone will not be included)

SECONDARY OUTCOMES:
Short-term (steroid-free) clinical response response to adalimumab in patients with moderate-to-severe ulcerative colitis | Week 8
  Short-term clinical response is defined as a decrease in the Mayo score of at least 3 points and at least 30 percent, with an accompanying decrease in the sub-score for rectal bleeding of at least 1 point or an absolute rectal-bleeding sub-score of 0 or 1
Short-term (steroid-free) clinical remission response to adalimumab in patients with moderate-to-severe ulcerative colitis | Week 8
  Short-term clinical remission is defined as a total Mayo score of 2 points or lower, with no individual sub-score exceeding 1 point
Short-term (steroid-free) clinical benefit to adalimumab in patients with moderate-to-severe ulcerative colitis | Week 8
  Short-term clinical benefit is defined as a meaningful clinical response with clear improvement in symptoms at discretion of the physician
Short-term (steroid-free) mucosal healing under adalimumab in patients with moderate-to-severe ulcerative colitis | Week 8
  Short-term mucosal healing is defined as a Mayo endoscopic sub-score of 0 or 1 at lower endoscopy performed between week 8 and 14
Short-term (steroid-free) complete mucosal healing under adalimumab in patients with moderate-to-severe ulcerative colitis | Week 8
  Short-term complete mucosal healing is defined as a Mayo endoscopic sub-score of 0 at lower endoscopy performed between week 8 and 14
Short-term (steroid-free) biological response to adalimumab in patients with moderate-to-severe ulcerative colitis | Week 8
  Short-term biological response is defined as a normalization of C-reactive protein (CRP) to <5 mg/L in patients with an elevated CRP at baseline (≥5 mg/L) and/or a normalization of faecal calprotectin to <250µg/g in patients with an elevated faecal calprotectin at baseline (≥250 µg/g)
Adalimumab dose-escalation free survival during adalimumab treatment | Through study completion, an average of 24 months
  Adalimumab dose-escalation free survival during adalimumab treatment
Adalimumab dose de-escalation free survival during adalimumab treatment | Through study completion, an average of 24 months
  Adalimumab dose de-escalation free survival during adalimumab treatment
Success of dose de-escalation within 6 months after dose de-escalation | Through study completion, an average of 24 months
  Success of dose de-escalation is defined as a persistent use of adalimumab at a dose of 40mg every other week for at least 6 months after dose de-escalation
Safety of adalimumab: Proportion of patients developing (serious) adverse events under adalimumab therapy during adalimumab treatment | Through study completion, an average of 24 months
  Proportion of patients developing (serious) adverse events under adalimumab therapy during adalimumab treatment
UC related hospitalization during adalimumab treatment | Through study completion, an average of 24 months
  Proportion of patient requiring ulcerative colitis related hospitalization during adalimumab treatment
UC related colectomy during follow-up | Through study completion, an average of 24 months
  Proportion of patient requiring colectomy during follow-up
Identification of variables associated with short-term outcome | Week 8
  Identifying variables associated with short-term outcome adalimumab
Identification of baseline variables associated with need for dose-escalation | Through study completion, an average of 24 months
  Identifying variables associated with need of dose escalation to adalimumab 40mg every week; variables to be evaluated will include sex, age, disease duration, familial history, extent of disease, previous medical therapy, concomitant medical therapy, adalimumab induction scheme, baseline serum values (Hb, albumin, CRP, ...), baseline endoscopic evaluation
Identification of baseline variables associated with successful dose-escalation | Through study completion, an average of 24 months
  Identifying variables associated with success of dose escalation to adalimumab 40mg every week; variables to be evaluated will include sex, age, disease duration, familial history, extent of disease, previous medical therapy, concomitant medical therapy, adalimumab induction scheme, baseline serum values (Hb, albumin, CRP, ...), baseline endoscopic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Marc Ferrante, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided